CLINICAL TRIAL: NCT02450058
Title: Fluorouracil, Epirubicin and Cyclophosphamide Versus Concurrent Epirubicin and Paclitaxel in Node Positive Early Breast Cancer Patients: a Randomized, Phase III Trial of Gruppo Oncologico Nord-Ovest - Mammella Intergruppo Group
Brief Title: Adjuvant FEC Versus EP in Breast Cancer (MIG5)
Acronym: MIG5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Principal Investigator, Lucia Del Mastro,MD, MD, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMI96.018
Record Dates: First submitted 2015-05-14; First posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer; Chemotherapy, Adjuvant
Keywords: early breast cancer; adjuvant chemotherapy; FEC; paclitaxel
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorouracil; Epirubicin; Cyclophosphamide; Paclitaxel

ARMS (2):
- FEC (Active Comparator): 5-Fluorouracil 600 mg/m2, epirubicin 60 mg/m2 and cyclophosphamide 600 mg/m2, intravenously on day 1, every 21 days
  Interventions: Drug: 5-fluorouracil; Drug: epirubicin; Drug: cyclophosphamide
- EP (Active Comparator): Epirubicin 90 mg/m2 and paclitaxel 175 mg/m2, 3-hour infusion on day 1, every 21 days
  Interventions: Drug: epirubicin; Drug: paclitaxel

INTERVENTIONS:
Drug: 5-fluorouracil — 600 mg/m2 intravenously on day 1, every 21 days for six cycles
  Arms: FEC
Drug: epirubicin — 60 mg/m2 intravenously on day 1, every 21 days for six cyles
  Arms: FEC
Drug: cyclophosphamide — 600 mg/m2, intravenously on day 1, every 21 days for six cycles
  Arms: FEC
Drug: epirubicin — 90 mg/m2 on day 1, every 21 days for four cycles
  Arms: EP
Drug: paclitaxel — 175 mg/m2, 3-hour infusion on day 1, every 21 days for four cycles
  Arms: EP

SUMMARY:
In this multicenter, randomized phase III trial, node positive early breast cancer patients are randomly assigned to receive either 6 cycles of FEC (5-fluorouracil 600 mg/m2, epirubicin 60 mg/m2 and cyclophosphamide 600 mg/m2, on day 1, every three weeks) or 4 cycles of EP (epirubicin 90 mg/m2 and paclitaxel 175 mg/m2, on day 1, every three weeks). The primary study endpoint is overall survival (OS). Secondary endpoints include toxicity and event free survival (EFS).

DETAILED DESCRIPTION:
At the time the Gruppo Oncologico Nord-Ovest- Mammella Intergruppo trial 5 (GONO-MIG5) was designed in 1996, paclitaxel was known to have efficacy in patients with advanced breast cancer, but its role was still to be established in the adjuvant setting. Therefore the GONO-MIG5 trial was designed to compare a standard anthracycline-containing chemotherapy regimen, i.e. 5fluorouracil, epirubicin, ciclophosphamide (FEC), given for 6 cycles to a new regimen containing both epirubicin and paclitaxel (EP), given concurrently, for 4 cycles. This latter regimen was chosen on the basis of the results obtained in metastatic breast cancer patients, where the combination of doxorubicin and paclitaxel was associated with more than 90% of objective response . Only four cycles of the new regimen were planned since the expected toxicity, particularly the cardiotoxicity, was high, and a short treatment duration was hoped to be the best strategy to obtain a favourable balance between the toxicity and the expected high efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically confirmed breast cancer who had undergone radical mastectomy or breast-conserving surgery in addition to full ipsilateral axillary lymph node dissection
* Lymph node-positive disease with less than 10 involved axillary lymph nodes
* Surgery performed not more than 5 weeks before randomization
* ECOG performance status 0
* Absolute neutrophil count ≥ 2,000/mm³
* WBC ≥ 3,000/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 1.5 times ULN
* Postoperative regional radiotherapy limited to the remaining breast admitted for patients who received breast-conserving surgery
* Written informed consent

Exclusion Criteria:

* Prior or concurrent ipsilateral or contralateral invasive breast carcinoma within the last 10 years
* Metastatic disease, including metastasis in the ipsilateral supraclavicular lymph nodes
* Prior chemotherapy or prior cytotoxic regimens or prior hormonal therapy
* Pregnant or nursing
* Other serious medical illness requiring medication, uncontrolled infections
* Other malignancy except adequately treated, cone-biopsied in situ carcinoma of the cervix or basal cell or squamous cell carcinoma of the skin
* Recent myocardial infarction, congestive heart failure, or serious arrhythmia

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1055 (Actual)
Dates: Start 1996-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
overall survival | within 11 years since the enrolment of the 1st patient
  estimated from the date of randomization to the date of death from any cause

SECONDARY OUTCOMES:
event free survival | within 11 years since the enrolment of the 1st patient
  from the date of randomization to the date of local recurrence, distant metastases, second primary cancer, or death from any cause
toxicity as measured according to the World Health Organization Criteria | within the first 30 days after the end of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Del Mastro, MD, Principal Investigator — IRCCS San Martino - IST, Istituto Nazionale per la Ricerca sul Cancro, Genoa
Locations (8):
- Italy (8):
  - Federico Castiglione, Alba
  - Ornella Garrone, Cuneo
  - Lucia Del Mastro, Genoa
  - Giovanna Cavazzini, Mantova
  - Andrea Michelotti, Pisa
  - Tiziana Scotto, Sassari
  - Antonio Durando, Torino
  - Saverio Danese, Torino